CLINICAL TRIAL: NCT05617911
Title: Clinical Comparison of Patellofemoral Pain Syndrome Outcomes After Blood Flow Restriction Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to lack of recruitment.
Sponsor: Gaylord Hospital, Inc (Other)
Collaborators: UConn Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202209SOK
Record Dates: First submitted 2022-11-01; First posted 2022-11-16 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Patellofemoral Pain Syndrome; Anterior Knee Pain Syndrome
Keywords: Blood Flow Restriction; Patellofemoral Pain Syndrome; Physical Therapy; Non-Specific Anterior Knee Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — salicylhydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Blood flow restriction and standard of care therapy (Experimental): The experimental BFR therapy will be incorporated into the standard therapy sessions and will not elongate the treatment session, quantity of sessions or incur any additional cost. As the participant progresses over time in therapy sessions, the discretion of the PT will determine when they have graduated beyond receiving any benefit from BFRT as demonstrated by quad strength.
  Interventions: Device: Blood Flow Restriction Cuff
- Sham and standard of care therapy (Placebo Comparator): The sham comparator control group will also follow the Exercise Protocol in their physical therapy sessions with a non inflated blood flow restriction cuff attached in the same position as the experimental group. Similar to the intervention group, as participant's progress in therapy, the Physical Therapist will use their clinical decision making to advance the person through resistance and repetition increases.
  Interventions: Procedure: Sham and standard of Care Therapy

INTERVENTIONS:
Device: Blood Flow Restriction Cuff — Blood Flow Restriction (BFR) involves the application of an external device to reduce arterial blood flow to the exercising area, while largely occluding venous return from that same area.
  Arms: Blood flow restriction and standard of care therapy
Procedure: Sham and standard of Care Therapy — SoC PT + non-inflated BFR cuff
  Arms: Sham and standard of care therapy

SUMMARY:
The purpose of this study is to determine if Blood Flow Restriction therapy improves patient related outcomes in those diagnosed with Patellofemoral Pain Syndrome compared to those in the sham comparator control group.

DETAILED DESCRIPTION:
Patellofemoral Pain Syndrome (PFPS), also known as Non-Specific Anterior Knee Pain (AKP), is a non-specific musculoskeletal condition characterized by loss of function and pain localized to the patella. PFPS affects up to 22% of the general population yearly, with females affected more so than males. Adolescents (28%, mixed gender) and elite athletes (up to 35% in knee dominant sports such as cycling) are also commonly affected, making this a relatively widespread condition. Additionally, PFPS has a generally unfavorable prognosis, with up to 40% of individuals failing conservative treatment after 1 year, and 57% reporting continued symptoms for 5 to 8-years following. Higher levels of baseline disability and longer duration of symptoms lead to an even poorer prognosis, making early recognition and novel treatments key. To complicate things further, the presence of negative psychosocial factors is commonly found in this population and may be a greater predictor of outcomes than physical ones.

Previously, biomechanical factors, such as maltracking of the patella and chondromalacia, have been called into question as potential causes of PFPS symptoms. However, both are now thought to be potential consequences of having PFPS. That being said, PFPS is generally accepted as a non-specific condition as there may be a number of different structures implicated as potential nociceptive drivers, and determining the exact tissue does not seem to be important to overall management strategies. This finding, in connection with the high prevalence of negative psychosocial factors, points less to a physiologically driven condition, and more towards a pain driven condition. While this theoretically makes diagnosing and treatment selection more ubiquitous, there does not seem to be a clear treatment strategy that works best for all patients. Despite a clear biomechanical cause, adjusting exercise selection or technique to include different loads and forces on the patella is still warranted based on patient presentation. For example, during open chain knee extension, the lowest loads are placed on the patella between 90- and 45-degree flexion, and open chain between 0 and 60 degrees. People with PFPS often benefit from adjusting the exercise selection, technique and load.

Recent research compared multiple different exercise strategies (combined core and hip work, knee work only, and open vs closed-chain), without any one program showing significant advantage over the others. A combination of these approaches may be best. One theme within PFPS exercise research that appears consistent is the high level of sensitivity and poor response to treatment where higher levels of pain are present. This is in contrast to tendon related pain, such as patellar tendinopathy, where working into moderate levels of pain seems to be helpful for outcomes.

The main mechanism driving improvements following exercise therapy for PFPS is not hypertrophy, but rather thought to be exercise induced hypoalgesia. This is a phenomenon where performing both acute bouts, as well as regular exercise (aerobic and resistance), reduces pain both in the short and long terms. Since exercise seems to reduce pain in both local and distant sites of the exercising area, it is thought to provide both local and systemic pain reducing effects. The magnitude and duration of the exercise seems to play an important role as well, with higher intensity and longer durations of exercising producing greater effects.

Since patients with PFPS are unable to achieve these desired parameters, alternative strategies need to be investigated. Two options may be blood flow restriction (BFR) therapy and low load training to failure, both of which may capture some of the hypoalgesic effects while minimizing AKP. BFR involves the application of an external device to reduce arterial blood flow to the exercising area, while largely occluding venous return from that same area. Exercise intensities generally range from 20-30% of the patients' 1 repetition maximum (1RM) weight, with relatively high repetitions (sometimes to failure); this is opposed to traditional resistance training at 70%+ of 1RM. BFR training has been demonstrated to amplify the effects of exercise induced hypoalgesia (in addition to a host of other physiological benefits) through unconfirmed mechanisms. Leading theories suggest that the lack of available oxygen to the exercising area may lead to: the activation of the endogenous opioid and cannabinoid systems; systemic changes to the cardiovascular system; or increased number of metabolites such as hydrogen ions and lactic acid, which may also be contributing factors.

Clinical research on the application of BFR in patients with PFPS has been both limited and mixed, with only two trials having been conducted in this area. One study from 2017 looked at high-load with BFR placebo, versus low-load BFR with leg press and knee extensions. Only the high-load group showed a modest medium-term effect on pain, lowering it for ~24 hours after BFR over the training period. The other paper from 2022 included both knee and hip strengthening exercises, comparing a low-load BFR group versus a high-load training group with no placebo; of note, the programs were not equated in terms of exercises completed. In this study, no significant difference was observed between groups. To date, there have been limited to no sham arms in studies where a BFR cuff was used. Given the potential for placebo effects, this was an important consideration in the design of the study.

Given the heterogeneity of these two studies, and the paucity of research in this area, the aim of the current study is to compare a low load training to failure (with BFR placebo) to low load BFR training to failure on the effect of pain related outcomes, function, strength and other measures. We hypothesize that BFR training will improve objective and subjective outcomes in patients with patellofemoral pain syndrome (PFPS) more than standard therapy with a sham BFR cuff.

Research aim 1: Determine whether the use of BFR improves patient-perceived function through a series of subjective patient-reported outcome measurements (PROs) throughout long-term recovery compared to patients in the sham control group. While we anticipate both groups may show improvement over time, we hypothesize that patients using BFR and the prescribed physical therapy protocol will demonstrate significantly improved PRO scores compared to the sham control group. These PROs include the Lower Extremity Functional Scale (LEFS), Knee Injury and Osteoarthritis Outcome Score for Patellofemoral Pain (KOOS-PF), the Single Assessment Numerical Evaluation (SANE), the Fear Avoidance Beliefs Questionnaire (FABQ), and Numerical Rating Scale (NRS) Pain Scale 1-10. Participants will be asked to complete PRO at the start of physical therapy (i.e. baseline), 4-weeks, 9-weeks or patient discharge if it is before the scheduled 9-week assessment, 6-month, and 12-month timepoints.

Research aim 2: Determine whether the use of BFR improves objective outcome measurements throughout prescribed physical therapy sessions compared to patients in the control group. While we anticipate both groups may show improvement over time, we hypothesize that patients using BFR and the prescribed physical therapy protocol will demonstrate significantly improved quadriceps isometric strength over the sham control group. Outcomes will be measured at the start of the physical therapy (i.e. baseline), 4-weeks, and 9-weeks or patient discharge if it is before the scheduled 9-week assessment.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of patellofemoral pain syndrome (PFPS) or non-specific anterior knee pain (NSAKP) and plan to attend Gaylord Specialty Healthcare Physical Therapy

Exclusion Criteria:

Member of a defined vulnerable population, women who are or suspected to be pregnant, prisoners, children under 15, or other protected populations

Body mass of the leg preventing the cuff from fitting properly

Radiographic evidence of osteoarthritis (≥ Kellgren-Lawrence Grade 2)

History of intra-articular injection into either knee within 3 -months

Uncontrolled or untreated inflammatory disorder

Acute inflammatory disorder

Uncontrolled Diabetes and/or peripheral neuropathy, impaired circulation

Uncontrolled cardiac conditions including uncontrolled hypertension

Areas of thrombophlebitis, thrombosis

Distal wounds or pain below the knee >4/10

History of or current rhabdomyolysis

Prolonged immobilization (>3 months)

Sickle cell anemia

Lymphadenectomy

Varicose veins, or a history of personal or immediate family history (parental or sibling) of deep vein thrombosis

Current infection at or below the level of cuff placement

Malignancies in or below the area to be treated

Other conditions/medications that would interfere with subject safety or data collection in the opinion of the PI

Subjects with an increased risk of non-response as determined by the therapist

Once entered in the study, a diagnosis change that affects participation

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sokolowski, Principal Investigator — Physical Therapist; Danielle Letendre, Principal Investigator — Physical Therapist
Locations (6):
- United States (6):
  - Gaylord Specialty Healthcare Outpatient Physical Therapy; Cheshire, Cheshire, Connecticut
  - Gaylord Specialty Healthcare Outpatient Physical Therapy; Cromwell, Cromwell, Connecticut
  - University of Connecticut Health Center, Farmington, Connecticut
  - Gaylord Specialty Healthcare Outpatient Physical Therapy; Madison, Madison, Connecticut
  - Gaylord Hospital, Wallingford, Connecticut
  - Gaylord Specialty Healthcare Outpatient Physical Therapy; Wallingford, Wallingford, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will become available to researchers that are interesting after analysis has been completed. Data will be available for 3 years after the date of completion.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available after analysis has been completed, and then will be available for 3 years after the date of completion.
Access Criteria: Qualified researchers will be allowed access to the deidentified data, and any other documents at the discretion of the primary investigators and research team

REFERENCES:
- [Background] Smith BE, Selfe J, Thacker D, Hendrick P, Bateman M, Moffatt F, Rathleff MS, Smith TO, Logan P. Incidence and prevalence of patellofemoral pain: A systematic review and meta-analysis. PLoS One. 2018 Jan 11;13(1):e0190892. doi: 10.1371/journal.pone.0190892. eCollection 2018. PMID 29324820
- [Background] Collins NJ, Bierma-Zeinstra SM, Crossley KM, van Linschoten RL, Vicenzino B, van Middelkoop M. Prognostic factors for patellofemoral pain: a multicentre observational analysis. Br J Sports Med. 2013 Mar;47(4):227-33. doi: 10.1136/bjsports-2012-091696. Epub 2012 Dec 13. PMID 23242955
- [Background] Lankhorst NE, van Middelkoop M, Crossley KM, Bierma-Zeinstra SM, Oei EH, Vicenzino B, Collins NJ. Factors that predict a poor outcome 5-8 years after the diagnosis of patellofemoral pain: a multicentre observational analysis. Br J Sports Med. 2016 Jul;50(14):881-6. doi: 10.1136/bjsports-2015-094664. Epub 2015 Oct 13. PMID 26463119
- [Background] Maclachlan LR, Matthews M, Hodges PW, Collins NJ, Vicenzino B. The psychological features of patellofemoral pain: a cross-sectional study. Scand J Pain. 2018 Apr 25;18(2):261-271. doi: 10.1515/sjpain-2018-0025. PMID 29794307
- [Background] Post WR, Dye SF. Patellofemoral Pain: An Enigma Explained by Homeostasis and Common Sense. Am J Orthop (Belle Mead NJ). 2017 Mar/Apr;46(2):92-100. PMID 28437494
- [Background] Saltychev M, Dutton RA, Laimi K, Beaupre GS, Virolainen P, Fredericson M. Effectiveness of conservative treatment for patellofemoral pain syndrome: A systematic review and meta-analysis. J Rehabil Med. 2018 May 8;50(5):393-401. doi: 10.2340/16501977-2295. PMID 29392329
- [Background] Powers CM, Ho KY, Chen YJ, Souza RB, Farrokhi S. Patellofemoral joint stress during weight-bearing and non-weight-bearing quadriceps exercises. J Orthop Sports Phys Ther. 2014 May;44(5):320-7. doi: 10.2519/jospt.2014.4936. Epub 2014 Mar 27. PMID 24673446
- [Background] Collins NJ, Barton CJ, van Middelkoop M, Callaghan MJ, Rathleff MS, Vicenzino BT, Davis IS, Powers CM, Macri EM, Hart HF, de Oliveira Silva D, Crossley KM. 2018 Consensus statement on exercise therapy and physical interventions (orthoses, taping and manual therapy) to treat patellofemoral pain: recommendations from the 5th International Patellofemoral Pain Research Retreat, Gold Coast, Australia, 2017. Br J Sports Med. 2018 Sep;52(18):1170-1178. doi: 10.1136/bjsports-2018-099397. Epub 2018 Jun 20. PMID 29925502
- [Background] Kountouris A, Cook J. Rehabilitation of Achilles and patellar tendinopathies. Best Pract Res Clin Rheumatol. 2007 Apr;21(2):295-316. doi: 10.1016/j.berh.2006.12.003. PMID 17512484
- [Background] Song JS, Spitz RW, Yamada Y, Bell ZW, Wong V, Abe T, Loenneke JP. Exercise-induced hypoalgesia and pain reduction following blood flow restriction: A brief review. Phys Ther Sport. 2021 Jul;50:89-96. doi: 10.1016/j.ptsp.2021.04.005. Epub 2021 Apr 23. PMID 33940556
- [Background] Misra G, Paris TA, Archer DB, Coombes SA. Dose-response effect of isometric force production on the perception of pain. PLoS One. 2014 Feb 4;9(2):e88105. doi: 10.1371/journal.pone.0088105. eCollection 2014. PMID 24505397
- [Background] Hughes L, Patterson SD. The effect of blood flow restriction exercise on exercise-induced hypoalgesia and endogenous opioid and endocannabinoid mechanisms of pain modulation. J Appl Physiol (1985). 2020 Apr 1;128(4):914-924. doi: 10.1152/japplphysiol.00768.2019. Epub 2020 Feb 27. PMID 32105522
- [Background] Giles L, Webster KE, McClelland J, Cook JL. Quadriceps strengthening with and without blood flow restriction in the treatment of patellofemoral pain: a double-blind randomised trial. Br J Sports Med. 2017 Dec;51(23):1688-1694. doi: 10.1136/bjsports-2016-096329. Epub 2017 May 12. PMID 28500081
- [Background] Constantinou A, Mamais I, Papathanasiou G, Lamnisos D, Stasinopoulos D. Comparing hip and knee focused exercises versus hip and knee focused exercises with the use of blood flow restriction training in adults with patellofemoral pain. Eur J Phys Rehabil Med. 2022 Apr;58(2):225-235. doi: 10.23736/S1973-9087.22.06691-6. Epub 2022 Jan 5. PMID 34985237
- [Background] Dolak KL, Silkman C, Medina McKeon J, Hosey RG, Lattermann C, Uhl TL. Hip strengthening prior to functional exercises reduces pain sooner than quadriceps strengthening in females with patellofemoral pain syndrome: a randomized clinical trial. J Orthop Sports Phys Ther. 2011 Aug;41(8):560-70. doi: 10.2519/jospt.2011.3499. Epub 2011 Jun 7. PMID 21654093
- [Background] Sisk D, Fredericson M. Update of Risk Factors, Diagnosis, and Management of Patellofemoral Pain. Curr Rev Musculoskelet Med. 2019 Dec;12(4):534-541. doi: 10.1007/s12178-019-09593-z. PMID 31773479
- [Background] Brightwell BD, Stone A, Li X, Hardy P, Thompson K, Noehren B, Jacobs C. Blood flow Restriction training After patellar INStability (BRAINS Trial). Trials. 2022 Jan 28;23(1):88. doi: 10.1186/s13063-022-06017-1. PMID 35090543
- [Background] Thiebaud RS, Yasuda T, Loenneke JP, Abe T. Effects of low-intensity concentric and eccentric exercise combined with blood flow restriction on indices of exercise-induced muscle damage. Interv Med Appl Sci. 2013 Jun;5(2):53-9. doi: 10.1556/IMAS.5.2013.2.1. Epub 2013 Jul 4. PMID 24265891

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Study terminated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Rating Scale: Enrollment
Description: The Numeric Pain Rating Scale is one question pain intensity scale that assesses the current, best, and worst pain level in the last 24 hours
Time Frame: This assessment will be collected upon enrollment in the study.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Numeric Pain Rating Scale: 1 Week
Description: as for outcome 1
Time Frame: This assessment will be collected 1-week into treatment
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Numeric Pain Rating Scale: 4 Weeks
Description: as for outcome 1
Time Frame: This assessment will be collected 4-weeks into treatment.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Numeric Pain Rating Scale: 9 Weeks/Discharge
Description: as for outcome 1
Time Frame: This assessment will be collected 9-weeks into treatment or at discharge, whatever comes first.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Numeric Pain Rating Scale: 6 Months
Description: as for outcome 1
Time Frame: This assessment will be collected 6 months post start date.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Numeric Pain Rating Scale: 12 Months
Description: as for outcome 1
Time Frame: This assessment will be collected 12 months post start date.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Lower Extremity Functional Scale: Enrollment
Description: The LEFS is a 20 question survey that is a valid PROM used for the measurement of lower extremity function based on the patients' initial function, ongoing progress, and long-term outcome
Time Frame: This assessment will be collected upon enrollment in the study.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Lower Extremity Functional Scale: 1 Week
Description: as for outcome 7
Time Frame: This assessment will be collected 1-week into treatment.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Lower Extremity Functional Scale: 4 Weeks
Description: as for outcome 7
Time Frame: This assessment will be collected 4-weeks into treatment.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Lower Extremity Functional Scale: 9 Weeks/Discharge
Description: as for outcome 7
Time Frame: This assessment will be collected 9-weeks into treatment or at discharge, whatever comes first.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Lower Extremity Functional Scale: 6 Months
Description: as for outcome 7
Time Frame: This assessment will be collected 6 months post start date.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

12. Primary Outcome: Lower Extremity Functional Scale: 12 Months
Description: as for outcome 7
Time Frame: This assessment will be collected 12 months post start date.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

13. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score for Patellofemoral Pain: Enrollment
Description: The KOOS-PF is an 11 question survey that is used to assess five outcomes; they include knee related Quality of Life, activities of daily living, sport and recreation function, activities, pain and symptoms
Time Frame: This assessment will be collected upon enrollment in the study.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

14. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score for Patellofemoral Pain: 1 Week
Description: as for outcome 13
Time Frame: This assessment will be collected1-week into treatment.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

15. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score for Patellofemoral Pain: 4 Weeks
Description: as for outcome 13
Time Frame: This assessment will be collected 4-weeks into treatment.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

16. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score for Patellofemoral Pain: 9 Weeks/Discharge
Description: as for outcome 13
Time Frame: This assessment will be collected 9-weeks into treatment or at discharge, whatever comes first.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

17. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score for Patellofemoral Pain: 6 Months
Description: as for outcome 13
Time Frame: This assessment will be collected 6 months post start date.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

18. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score for Patellofemoral Pain: 12 Months
Description: as for outcome 13
Time Frame: This assessment will be collected 12 months post start date.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

19. Primary Outcome: Single Assessment Numerical Evaluation: Enrollment
Description: The SANE is a two item questionnaire used globally to assess function
Time Frame: This assessment will be collected upon enrollment in the study.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

20. Primary Outcome: Single Assessment Numerical Evaluation: 1 Week
Description: The SANE is a two item questionnaire used globally to assess function
Time Frame: This assessment will be collected 1-week into treatment.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

21. Primary Outcome: Single Assessment Numerical Evaluation: 4 Weeks
Description: The SANE is a two item questionnaire used globally to assess function
Time Frame: This assessment will be collected 4-weeks into treatment.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

22. Primary Outcome: Single Assessment Numerical Evaluation: 9 Weeks/Discharge
Description: The SANE is a two item questionnaire used globally to assess function
Time Frame: This assessment will be collected 9-weeks into treatment or at discharge, whatever comes first.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

23. Primary Outcome: Single Assessment Numerical Evaluation: 6 Months
Description: The SANE is a two item questionnaire used globally to assess function
Time Frame: This assessment will be collected 6 months post start date.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

24. Primary Outcome: Single Assessment Numerical Evaluation: 12 Months
Description: The SANE is a two item questionnaire used globally to assess function
Time Frame: This assessment will be collected 12 months post start date.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

25. Primary Outcome: Tenger Activity Scale: Enrollment
Description: The Tenger Activity Scale aims to provide a standardized method in determining the level of activity prior to injury and level of activity post injury that can be documented on a numerical scale.
Time Frame: This assessment will be collected upon enrollment.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

26. Primary Outcome: Tenger Activity Scale: 6 Months
Description: as for outcome 25
Time Frame: This assessment will be collected 6 months post start date.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

27. Primary Outcome: Tenger Activity Scale: 12 Months
Description: as for outcome 25
Time Frame: This assessment will be collected 12 months post start date.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

28. Primary Outcome: Fear Avoidance Beliefs Questionnaire: Enrollment
Description: The Fear Avoidance Belief Questionnaire is a 16 question likert scale questionnaire aimed at assessing how everyday activities assess the patient's current level of pain
Time Frame: This assessment will be collected upon enrollment in the study.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

29. Primary Outcome: Fear Avoidance Beliefs Questionnaire: 1 Week
Description: as for outcome 28
Time Frame: This assessment will be collected 1-week into treatment.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

30. Primary Outcome: Fear Avoidance Beliefs Questionnaire: 4 Weeks
Description: as for outcome 28
Time Frame: This assessment will be collected 4-weeks into treatment.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

31. Primary Outcome: Fear Avoidance Beliefs Questionnaire: 9 Weeks/Discharge
Description: as for outcome 28
Time Frame: This assessment will be collected 9-weeks into treatment or at discharge, whatever comes first.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

32. Primary Outcome: Fear Avoidance Beliefs Questionnaire: 6 Months
Description: as for outcome 28
Time Frame: This assessment will be collected 6 months post start date.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

33. Primary Outcome: Fear Avoidance Beliefs Questionnaire: 12 Months
Description: as for outcome 28
Time Frame: This assessment will be collected 12 months post start date.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Quadricep Isometric Strength: Enrollment
Description: Quadricep Isometric Strength is the amount of strength shown in a patient's quadricep muscle via isometric dynomometry
Time Frame: This assessment will be collected upon enrollment in the study.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Quadricep Isometric Strength: 1 Week
Description: Quadricep Isometric Strength is the amount of strength shown in a patient's quadricep muscle via isometric dynomometry
Time Frame: This assessment will be collected 1-week into treatment.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: Quadricep Isometric Strength: 4 Weeks
Description: Quadricep Isometric Strength is the amount of strength shown in a patient's quadricep muscle via isometric dynomometry
Time Frame: This assessment will be collected 4-weeks into treatment.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

37. Secondary Outcome: Quadricep Isometric Strength: 9 Weeks/Discharge
Description: Quadricep Isometric Strength is the amount of strength shown in a patient's quadricep muscle via isometric dynomometry
Time Frame: This assessment will be collected 9-weeks into treatment or at discharge, whatever comes first.
Population: Study terminated and participant withdrawal
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 participant withdrew, no participants were monitored/assessed for adverse events
Description: Descriptions of adverse events and/or serious adverse events do not differ from clinicaltrials.gov definitions.
Arm/Group | Blood Flow Restriction and Standard of Care Therapy | Sham and Standard of Care Therapy
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT05617911/Prot_SAP_001.pdf